CLINICAL TRIAL: NCT04047381
Title: Validity and Reliability of the Turkish Version of Atrial Fibrillation Impact Questionnaire (AFImpact)
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assistant Professor, Bezmialem Vakif University
Other Study IDs: bvumzeren03
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Quality of life
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Turkish patients diagnosed with atrial fibrillation
  Interventions: Other: Measurement of Quality of Life

INTERVENTIONS:
Other: Measurement of Quality of Life — Quality of life will be measured using Atrial Fibrillation Impact Questionnaire, Short Form-36 and Pittsburgh Sleep Quality Index

SUMMARY:
Validity and reliability of the Turkish version of 'Atrial Fibrillation Impact Questionnaire (AFImpact)' will be evaluated in the study.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia with a reported incidence of 2.1% in Turkish population aged 60 and above. Although a minority of patients have minimal or no symptoms, palpitations, dyspnea and fatigue are frequently reported by AF patients. It is well documented that AF patients, including those with no symptoms, have poorer quality of life (QoL) compared to healthy population. Worrying about their condition, side effects of treatments and worsening health are the other factors that have an impact on QoL, beside symptoms. Management of QoL is a key therapeutic goal in AF treatment and guidelines recommend that QoL in these patients should be measured regularly. There is a concern in the literature that generic QoL measures may not be sufficiently sensitive or specific to measure AF related QoL, thus using disease specific QoL measures are recommended for AF patients. An AF-specific quality of life measure is lacking in Turkish language, thus our aim in this study is to validate the Turkish version of 'Atrial Fibrillation Impact Questionnaire (AFImpact)' in Turkish AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paroxysmal, persistant or permanent atrial fibrillation
* To be able to read and understand Turkish

Exclusion Criteria:

* Diagnosis of heart failure or any chronic lung diseases
* Recent coronary bypass surgery
* Previous heart valve surgery
* Rheumatic valvular heart disease
* Recent acute myocardial infarction
* Having a pacemaker

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish patients diagnosed with atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Impact Questionnaire (AFImpact) | 5 minutes
  AFImpact is a 18-item disease specific questionnaire that enables respondents to recall how often their atrial fibrillation affected their lives over the past seven days. Each item is scored on a seven-point likert scale (between 0 and 6 point, 6 point is being the most frequent). Higher scores indicate poorer quality of life.

SECONDARY OUTCOMES:
Short-form 36 (SF-36) | 10 minutes
  SF-36 is a generic quality of life questionnaire that is widely used in clinical research. It consists of 36 items and yields an 8-scale profile of functional health and well-being scores as well as two summary scores of physical and mental health. A higher score on a 0-100 scale indicates a better quality of life.
Pittsburgh Sleep Quality Index | 5 minutes
  Pittsburgh Sleep Quality Index is a 24-item questionnaire that assess subjective sleep quality over the past month. It consists of seven clinical domains which are also pooled linearly to get a global score.Each item is scored on a 0-3 likert scale and higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Institute of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided